CLINICAL TRIAL: NCT06481306
Title: A Phase 1/2a, First-in-human, Randomized, Double-blinded, Placebo-controlled, Dose-finding Study in Healthy Volunteers and Participants With Sickle Cell Disease to Evaluate the Safety and Tolerability, Pharmacokinetics, Pharmacodynamics, pH and Food Effect, and Preliminary Efficacy of BMS-986470
Brief Title: A Study to Evaluate BMS-986470 in Healthy Volunteers and Participants With Sickle Cell Disease
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA230-1019; 2023-510283-12 (Other: EU CTR); U1111-1301-6753 (Other: WHO)
Record Dates: First submitted 2024-06-25; First posted 2024-07-01 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2026-01

CONDITIONS: Anemia, Sickle Cell; Healthy Volunteers
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Famotidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort A Part 1 (Experimental)
  Interventions: Drug: BMS-986470; Drug: Placebo
- Cohort A Part 2 (Experimental)
  Interventions: Drug: BMS-986470; Drug: Placebo
- Cohort A Part 3 (Experimental)
  Interventions: Drug: BMS-986470; Drug: Famotidine
- Cohort B Part 1 (Experimental)
  Interventions: Drug: BMS-986470; Drug: Placebo
- Cohort B Part 2 (Experimental)
  Interventions: Drug: BMS-986470

INTERVENTIONS:
Drug: BMS-986470 — Specified dose on specified days
Drug: Placebo — Specified dose on specified days
  Arms: Cohort A Part 1; Cohort A Part 2; Cohort B Part 1
Drug: Famotidine — Specified dose on specified days
  Arms: Cohort A Part 3

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability, pharmacokinetics and pharmacodynamics, pH and food effect, and preliminary efficacy of BMS-986470 in healthy volunteers and participants with sickle cell disease.

ELIGIBILITY:
Inclusion Criteria

- Cohort A.

i) Healthy male and female (who are not of childbearing potential) participants, as determined by the investigator based on medical history and other determinations. Females not of childbearing potential must have been amenorrhoeic for at least 12 months without an alternative medical cause and have follicle-stimulating hormone (FSH) levels of at least 40 IU/L or have undergone a hysterectomy, bilateral oophorectomy, or bilateral salpingectomy.

ii) Body mass index (BMI) of 18.0 to 32.0 kg/m^2, inclusive. BMI = weight (kg)/ (height [m])^2 as measured at screening.

iii) No evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG, or clinical laboratory assessments beyond what is consistent with the target population.

- Cohort B.

i) Participants with a documented diagnosis of Sickle Cell Disease (SCD) with genotype HbSS, HbSβ0-thal, or HbSβ+-thal.

ii) Participants with ≥ 4 vaso-occlusive crises (VOCs) within the previous 12 months or ≥ 2 VOCs within the previous 6 months.

iii) Participant has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

iv) Must have the following laboratory values:.

A. Hemoglobin ≥ 5.5 and ≤ 12 g/dL (males) or ≥ 5.5 and ≤ 10.6 g/dL (females).

B. Absolute neutrophil count ≥ 1500/μL.

C. Platelet count ≥ 100 × 10^3/μL.

D. Absolute reticulocyte count > 100 × 10^3/μL or > 50 × 10^3/μL if taking hydroxyurea.

Exclusion Criteria

- Cohort A.

i) Any significant medical condition or any condition that confounds the ability to interpret data from the study.

ii) Participant has any condition, including the presence of laboratory abnormalities, that places the participant at unacceptable risk if the participant was to participate in the study.

iii) Any major surgery or planned surgery (except GI surgery) within 12 weeks of the first study intervention administration.

- Cohort B.

i) Participants with any condition, including significant acute or chronic medical illness, active or uncontrolled infection, or the presence of laboratory abnormalities, that places participants at unacceptable risk if participating in this study.

ii) Participants with more than 6 severe VOCs defined as VOCs requiring ≥ 24 hours of hospital admission within 12 months prior to the first dose of study intervention or any VOC requiring ≥ 24 hours of hospital admission within 30 days prior to the first dose of study intervention.

iii) Participants with any episode of acute chest syndrome within the last 6 months prior to the first dose of study intervention.

iv) Creatinine clearance (CrCl) < 60 mL/min/1.72m2 using Chronic Kidney Disease Epidemiology (CKD-EPI) equation

* Cohort A and B.

  i) Participant is receiving regularly scheduled RBC or platelet transfusions or has received a RBC transfusion within 28 days and a platelet transfusion within 14 days prior to starting treatment with BMS-986470.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2027-01-06 (Estimated); Study Completion 2027-11-16 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to 26 months
Number of participants with serious adverse events (SAEs) | Up to 26 months
Number of participants with AEs meeting protocol-defined Dose Limiting Toxicity (DLT) criteria | Up to 26 months
Number of participants with AEs leading to discontinuation | Up to 26 months
Number of deaths | Up to 26 months

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to Day 28
  Cohort A Parts 1 and 2 and Cohort B Part 1
Area under the concentration-time curve (AUC) | Up to Day 28
  Cohort A Parts 1 and 2 and Cohort B Part 1
Time of maximum observed plasma concentration (Tmax) | Up to Day 28
  Cohort A Parts 1 and 2 and Cohort B Part 1
Dose proportionality of BMS-986470 for Cmax and AUC | Up to Day 28
  Assessed by using the slope of a statistical linear relationship between the ln-transformed PK parameters AUC and Cmax and the ln-transformed dose will be fitted by using power model
Change from baseline in total hemoglobin (Hb) | Up to 26 months
  Cohort A Part 2, Cohort B Parts 1 and 2
Change from baseline in total Hb fractions: adult Hb (HbA) | Up to Day 28
  Cohort A Part 2
Change from baseline in total Hb fractions: fetal Hb (HbF) | Up to 26 months
  Cohort A Part 2, Cohort B Parts 1 and 2
Change from baseline in total Hb fractions: sickle Hb (HbS) | Up to 26 months
  Cohort B
Change from baseline in markers of red blood cell (RBC) lysis: total Hb | Up to 26 months
  Cohort B
Change from baseline in markers of RBC lysis: aspartate aminotransferase (AST) | Up to 26 months
  Cohort B
Change from baseline in markers of RBC lysis: lactate dehydrogenase (LDH) | Up to 26 months
  Cohort B
Change from baseline in markers of RBC lysis: total bilirubin | Up to 26 months
  Cohort B
Change from baseline in markers of RBC lysis: indirect bilirubin | Up to 26 months
  Cohort B
Change from baseline in markers of RBC lysis: haptoglobin | Up to 26 months
  Cohort B
Change from baseline in markers of RBC lysis: absolute reticulocyte count | Up to 26 months
  Cohort B
Change from baseline in markers of RBC lysis: reticulocyte percentage of RBCs | Up to 26 months
  Cohort B
Number of participants achieving HbF ≥ 10% | Up to 26 months
  Cohort B
Number of participants achieving HbF ≥ 20% | Up to 26 months
  Cohort B
Number of participants achieving HbF ≥ 30% | Up to 26 months
  Cohort B

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (19):
- United States (13):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California San Diego - La Jolla, La Jolla, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Yale-New Haven Hospital, New Haven, Connecticut
  - Local Institution - 0017, Atlanta, Georgia
  - Local Institution - 0034, Chicago, Illinois
  - Local Institution - 0001, Lenexa, Kansas
  - Local Institution - 0024, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Thomas Jefferson University - Medicine/GI and Hepatology, Philadelphia, Pennsylvania
  - Local Institution - 0032, Pittsburgh, Pennsylvania
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Virginia Commonwealth University (VCU) Medical Center, Richmond, Virginia
- France (3):
  - Institut de cancérologie Strasbourg Europe (ICANS), Strasbourg, Alsace
  - Assistance Publique Hôpitaux de Marseille - Hôpital de la Timone, Marseille
  - Hôpital Universitaire Necker Enfants Malades, Paris
- United Kingdom (3):
  - University Hospitals Sussex NHS Foundation Trust, East Sussex, Brighton And Hove
  - King's College Hospital, London, London, City of
  - Local Institution - 0005, Leeds

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria.
  Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at:
  https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06481306.html